CLINICAL TRIAL: NCT02800135
Title: Performance of Diuretic Stress Test in Predicting Short Term Renal Recovery in Oliguric Critically-ill Patients
Brief Title: Performance of Diuretic Stress Test in Predicting Short Term Renal Recovery in Oliguric Critically-ill Patients Recovery in the Short Term
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: departure of the coordinating investigator from another institution
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1408024; 141521A-11 (Other: ANSM); 2014-005146-22 (EudraCT Number)
Record Dates: First submitted 2015-12-18; First posted 2016-06-15 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Critical Illness; Oliguria
MeSH Terms: conditions — Critical Illness; Oliguria | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Furosemide stress test (Experimental)
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Furosemide — 1.0 mg/kg of intravenous furosemide. In order to minimize the risk of hypovolemia, urine output will be replaced ml for ml with either Ringers lactate or normal saline for six hours after the furosemide stress test.

SUMMARY:
Acute kidney injury (AKI) is a common disorder and associated with high morbidity and mortality. However, distinguishing transient AKI from persistent AKI may help in individualizing treatment and limit short and long term consequences of AKI. Previous studies suggested usual urinary indices to perform poorly for separating transient from persistent AKI in an unselected population of critically ill patients. The recent KDIGO (Kidney Disease Improving Global Outcomes) guidelines underlined the need for additional strategies in estimating renal short term prognosis.

Recently, a Furosemide stress test (FST) was validated in a cohort of unselected critically ill patients. This stress test performance was found to be good in predicting capacity to identify those patients that will progress to advanced stage AKI. Additionally, FST performance was higher than those of usual renal biomarker. The limited sample size of this preliminary study however precluded adjustment for usual confounders including oliguria.

The primary objective of this study is to assess diagnostic performance of FST in differentiating transient and persistent AKI. Secondary objectives are to assess diagnostic performance of FST in predicting need for renal replacement therapy, and to confirm FST results after adjustment for confounders.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18 y.o)
* AKI stage 1 or more according to KDIGO
* Oliguria as defined by an oliguria lower than 0.5 mL/Kg
* Affiliation to the National Medical Insurance

Exclusion Criteria:

* Pregnancy
* Chronic kidney disease stage 4 or more
* Need for fluid bolus (>1000 mL crystalloids or equivalent) or need for vasopressors increases or introduction in the 2 hours preceding inclusion
* Evidence of obstructive renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
Number of patients with renal recovery | day 3

SECONDARY OUTCOMES:
natriuresis(mmol/L) | day 0 to day 3
fractional excretion of sodium(%) | day 0 to day 3
fractional excretion of urea (%), | day 0 to day 3
U/P urea ratio(mg.dl-1/ mg.dl-1) | day 0 to day 3
U/P creatinine ratio (mg.dl-1/ mg.dl-1) | day 0 to day 3

CONTACTS AND LOCATIONS:
Overall Officials: Michael DARMON, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (4):
- France (4):
  - CHU de CLERMONT-FERRAND, Clermont-Ferrand
  - CHU de MONTPELLIER, Montpellier
  - CHU de SAINT-ETIENNE, Saint-Etienne
  - CHRU de STRASBOURG, Strasbourg

IPD SHARING:
Plan to Share IPD: No